CLINICAL TRIAL: NCT01027585
Title: Effects of Cinnamon on Postprandial Blood Glucose, and Insulin in Subjects With Type 2 Diabetes or Impaired Glucose Tolerance
Brief Title: The Effects of Cinnamon on Postprandial Blood Glucose, and Insulin in Subjects With Impaired Glucose Tolerance
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Lars Stavenow, Departments of Medicine, Malmö University Hospital
Other Study IDs: 353/2008a
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To study the effect of cinnamon on postprandial blood glucose, and plasma concentrations of insulin in subjects with impaired glucose tolerance.

DETAILED DESCRIPTION:
Ten subjects with impaired glucose tolerance were assessed in a crossover trial. A standard 75 g oral glucose tolerance test (OGTT) was served with placebo or cinnamon capsules. Finger-prick capillary and venous blood samples were taken before and 15, 30, 45, 60, 90, 120, 150, and 180 min after the start of the OGTT to measure glucose, and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients were selected for the study on the basis of the following inclusion criteria: diagnosis of impaired glucose tolerance for < 12 months before enrollment. Glucose tolerance status and fasting blood glucose levels were evaluated using the criteria established by the American Diabetes Association.

Exclusion Criteria:

* Subjects who had thyroid disorders, or used insulin, oral hypoglycemics, and insulin-sensitizing drugs within 60 days before enrollment were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects were recruited from the population in southern Sweden.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-05; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Hlebowicz, MD, PhD, Principal Investigator — Skane University Hospital